CLINICAL TRIAL: NCT01294345
Title: Personalized Genomic Research
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110093; 11-HG-0093
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Genetics; Genetic Disease; Genetic Linkage; Birth Defects; Genetic Variation
Keywords: Genomics; Personalized; Congenital Malformations; Birth Defects
MeSH Terms: conditions — Genetic Diseases, Inborn; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biospecimens include blood and tissue samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- personalized genomics: genetic/genomic syndromes

SUMMARY:
Background:

- Congenital malformations, sometimes called birth defects, occur because of a difference in early human development. There are many different types of congenital malformations, and some of these can be caused by changes in genetic material. Researchers are interested in studying individuals with these congenital malformations to better understand the causes and the effects of certain congenital malformations.

Objectives:

* To understand more about what causes congenital malformations that arise in early human development.
* To learn if genetic causes can be found to explain why a person has a congenital malformation.

Eligibility:

- Individuals who have been diagnosed with a congenital malformation.

Design:

* Participants will be seen at the National Institutes of Health for a series of visits over 3 to 4 days. Participants will be asked to provide copies of past medical records and test results for review, and will be asked questions about pregnancy/prenatal history, birth, newborn, medical, developmental, and family history.
* Parents or siblings of participants may also be asked to provide information for research purposes.
* Participants may have additional medical evaluations as part of this study, including any of the following tests:
* Physical examinations
* Other consultations as clinically indicated
* Blood samples for genetic testing
* Tissue biopsy for genetic testing
* Photographs of affected areas, such as front and side views of the face and other body parts that may be involved in a congenital malformation, like the hands and feet.
* Other tests as indicated by a specific malformation, such as organ ultrasounds.
* No additional invasive testing, testing requiring sedation, or testing involving radiation is planned for this protocol. These tests, if performed, would involve a separate consent....

DETAILED DESCRIPTION:
Recent advances in genomic techniques are making possible a new wave of genetic discovery. We hope to couple genomic techniques with more traditional methods involved in genetic discovery in order to investigate a broad range of conditions for which there is strong evidence that genetic factors are involved. To accomplish this, we plan to enroll approximately five families, in whom members have congenital malformations consistent with an error of early human development, in our research protocol each year. Patients will be referred from outside clinicians or may self-refer, and may be seen at the NIH Clinical Center or may send samples for testing. Some participants, for whom we already have DNA or tissue stored, may be reconsented for specific participation in this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:
* For affected individuals (individuals who are related to a person who meets criteria (1) below may also be included in the research protocol), determination of clinical criteria for inclusion will be determined by prior medical record review before participation.
* Presence of a congenital malformation or related medical finding thought to be related to errors in early human development.

EXCLUSION CRITERIA:

* Anyone unwilling to provide informed consent (for themselves as adults, or on behalf of their children as minors, or on behalf of an adult who is unable to provide consent for themselves) or assent.
* Clear evidence for the presence of a condition for which diagnostic testing is already available.

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study populations are from hospital and clinical settings.
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2011-01-24 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Natural history | lifetime
  genomic diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Kruszka, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kruszka P, Porras AR, Addissie YA, Moresco A, Medrano S, Mok GTK, Leung GKC, Tekendo-Ngongang C, Uwineza A, Thong MK, Muthukumarasamy P, Honey E, Ekure EN, Sokunbi OJ, Kalu N, Jones KL, Kaplan JD, Abdul-Rahman OA, Vincent LM, Love A, Belhassan K, Ouldim K, El Bouchikhi I, Shukla A, Girisha KM, Patil SJ, Sirisena ND, Dissanayake VHW, Paththinige CS, Mishra R, Klein-Zighelboim E, Gallardo Jugo BE, Chavez Pastor M, Abarca-Barriga HH, Skinner SA, Prijoles EJ, Badoe E, Gill AD, Shotelersuk V, Smpokou P, Kisling MS, Ferreira CR, Mutesa L, Megarbane A, Kline AD, Kimball A, Okello E, Lwabi P, Aliku T, Tenywa E, Boonchooduang N, Tanpaiboon P, Richieri-Costa A, Wonkam A, Chung BHY, Stevenson RE, Summar M, Mandal K, Phadke SR, Obregon MG, Linguraru MG, Muenke M. Noonan syndrome in diverse populations. Am J Med Genet A. 2017 Sep;173(9):2323-2334. doi: 10.1002/ajmg.a.38362. Epub 2017 Jul 27. PMID 28748642
- [Background] Weiss K, Wigby K, Fannemel M, Henderson LB, Beck N, Ghali N, Study DDD, Anderlid BM, Lundin J, Hamosh A, Jones MC, Ghedia S, Muenke M, Kruszka P. Haploinsufficiency of ZNF462 is associated with craniofacial anomalies, corpus callosum dysgenesis, ptosis, and developmental delay. Eur J Hum Genet. 2017 Aug;25(8):946-951. doi: 10.1038/ejhg.2017.86. Epub 2017 May 17. PMID 28513610
- [Derived] Murdock DR, Donovan FX, Chandrasekharappa SC, Banks N, Bondy C, Muenke M, Kruszka P. Whole-Exome Sequencing for Diagnosis of Turner Syndrome: Toward Next-Generation Sequencing and Newborn Screening. J Clin Endocrinol Metab. 2017 May 1;102(5):1529-1537. doi: 10.1210/jc.2016-3414. PMID 28324009
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-HG-0093.html